CLINICAL TRIAL: NCT03394768
Title: An Observational Study Comparing NICOM-Cheetah Versus Flotrac-Vigileo for Cardiac Output Monitoring in the Surgical Intensive Care Unit.
Brief Title: Comparison Between NICOM-Cheetah and Flotrac-Vigileo for Cardiac Output Monitoring.
Status: Terminated | Type: Observational
Why Stopped: Interim analysis shown futility to continue due to lack of benefit.
Sponsor: Changi General Hospital (Other)
Responsible Party: Principal Investigator, Chang See Seong, Consultant, Changi General Hospital
Other Study IDs: 2017/2820; CHF2017.08-S (Other Grant/Funding Number: CGH Research Grant 2017)
Record Dates: First submitted 2018-01-03; First posted 2018-01-09 (Actual); Results first posted 2021-03-03 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Cardiac Output, Low
MeSH Terms: conditions — Cardiac Output, Low

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- NICOM Cheetah®: Patients will be treated as per department protocols and no additional intervention will be performed. Each patient will have an arterial catheter inserted as per our usual practice. All patients will have the FloTrac® connected to the arterial catheter (standard of care in CGH SICU) and the NICOM Cheetah® electrodes placed on the skin across the anterior thoracic wall. The NICOM CO monitor involves the application of non-invasive sensor strips. In this study, it will be applied to patients receiving the FloTrac (standard of care), on top of the standard care of monitoring with Flotrac.
  Interventions: Other: No additional intervention
- FloTrac®: Same patient population as the NICOM Cheetah® group as described above as all patients will have the FloTrac® connected to the arterial catheter (standard of care in CGH SICU) and the NICOM Cheetah® electrodes placed on the skin across the anterior thoracic wall. The FloTrac CO monitor is the current standard of care for cardiac output monitoring in the SICU of CGH. All patients deemed to require cardiac output monitoring will receive the FloTrac (as per departmental practice).
  Interventions: Other: No additional intervention

INTERVENTIONS:
Other: No additional intervention — Patients will be treated as per department protocols and no additional intervention will be performed

SUMMARY:
Cardiac output (CO) monitoring is an important tool in critically ill patients with haemodynamic instability. Traditionally, this has been accomplished using the pulmonary artery catheter (PAC). However, its use has been associated with various complications such as pneumothorax, arrhythmia, infection, pulmonary valve injury and embolism. This has led to the development of various minimally invasive cardiac output monitoring devices such as the oesophageal Doppler, PiCCO®, NiCCO® and FloTrac®. These devices however have their inherent limitations and though minimally invasive, are still not without risks to the patient. More recently a completely non-invasive CO monitoring device, NICOM Cheetah® has been introduced. Its use is based on thoracic bioreactance and it involves placement of 4 electrodes on either side of the thorax and it analyses changes in the phase of electrical voltage signal to the current applied across the thorax. Initial validation studies on the NICOM Cheetah® device revealed promising results. This study intends to compare cardiac output monitoring capabilities of the NICOM Cheetah® device using the FloTrac® CO monitor as a reference.

DETAILED DESCRIPTION:
This will be a single centre prospective observational study. 50 consecutive patients admitted to the surgical intensive care unit (SICU) who are deemed to require cardiac output monitoring by the treating intensivist will be studied. Data collection is planned to be carried out over 2 consecutive years. Inclusion criteria are: 1) Patients who are deemed to require cardiac output monitoring. 2) Patients 21 years old and above. 3) American Society of Anesthesiologist (ASA) physical status 1 to 4. Exclusion criteria are: 1) Patients who are not on mechanical ventilation. 2) Patients who are not in sinus rhythm. 3) Patients with allergy to adhesive tapes. Patients will be treated as per department protocols and no additional intervention will be performed. Each patient will have an arterial catheter inserted as per our usual practice. All patients will have the FloTrac® connected to the arterial catheter (standard of care in CGH SICU) and the NICOM Cheetah® electrodes placed on the skin across the anterior thoracic wall. The FloTrac CO monitor is the current standard of care for cardiac output monitoring in the SICU of CGH. All patients deemed to require cardiac output monitoring will receive the FloTrac (as per departmental practice). The NICOM CO monitor involves the application of non-invasive sensor strips. In this study, it will be applied to patients receiving the FloTrac (standard of care), on top of the standard care of monitoring with Flotrac. For each patient, standard demographic and SICU data (age, gender, comorbidities, ASA score, admission diagnosis, type of surgery, cause of haemodynamic instability, mean arterial pressure (MAP) and central venous pressure (CVP) at the time of instituting cardiac output (CO) monitoring, use of inotropic support, presence of renal replacement therapy, presence of mechanical ventilation and APACHE II score) will be collected. Cardiac Index (CI) values simultaneously recorded by the NICOM Cheetah® and FloTrac® on a 15-minutely basis for the first 10-hour period will also be collected. These data will be automatically recorded by the FloTrac® Vigilance monitor and the Cheetah NICOM monitor and transcribed to a data entering/analysis software by the principal and co-principal investigators for data analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are deemed to require cardiac output monitoring.
* Patients 21 years old and above
* American Society of Anesthesiologist (ASA) physical status 1 to 4

Exclusion Criteria:

* Patients who are not on mechanical ventilation.
* Patients who are not in sinus rhythm.
* Patients with allergy to adhesive tapes

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the surgical intensive care unit (SICU) who are deemed to require cardiac output monitoring by the treating intensivist
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2018-08-10 (Actual); Primary Completion 2021-01-05 (Actual); Study Completion 2021-01-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: See Seong Chang, MBBS, MMed, Principal Investigator — Changi General Hospital; Louis Ng, MBBS, ANZCA, Principal Investigator — Changi General Hospital
Locations (1):
- Surgical Intensive Care Unit, Changi General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
IPD will not be available to anyone else other than the investigators of this study

REFERENCES:
- [Background] Squara P, Denjean D, Estagnasie P, Brusset A, Dib JC, Dubois C. Noninvasive cardiac output monitoring (NICOM): a clinical validation. Intensive Care Med. 2007 Jul;33(7):1191-1194. doi: 10.1007/s00134-007-0640-0. Epub 2007 Apr 26. PMID 17458538
- [Background] Raval NY, Squara P, Cleman M, Yalamanchili K, Winklmaier M, Burkhoff D. Multicenter evaluation of noninvasive cardiac output measurement by bioreactance technique. J Clin Monit Comput. 2008 Apr;22(2):113-9. doi: 10.1007/s10877-008-9112-5. Epub 2008 Mar 14. PMID 18340540
- [Background] Marque S, Cariou A, Chiche JD, Squara P. Comparison between Flotrac-Vigileo and Bioreactance, a totally noninvasive method for cardiac output monitoring. Crit Care. 2009;13(3):R73. doi: 10.1186/cc7884. Epub 2009 May 19. PMID 19454009
- [Background] Mehta Y, Arora D. Newer methods of cardiac output monitoring. World J Cardiol. 2014 Sep 26;6(9):1022-9. doi: 10.4330/wjc.v6.i9.1022. PMID 25276302

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants recruited from the surgical intensive care unit of Changi General Hospital, Singapore, from 2018 until 2021
Groups:
- All Participants: Patients will be treated as per department protocols and no additional intervention will be performed. Each patient will have an arterial catheter inserted as per our usual practice. All patients will have the FloTrac® connected to the arterial catheter (standard of care in CGH SICU) and the NICOM Cheetah® electrodes placed on the skin across the anterior thoracic wall. The NICOM CO monitor involves the application of non-invasive sensor strips. In this study, it will be applied to patients receiving the FloTrac (standard of care), on top of the standard care of monitoring with Flotrac.
  No additional intervention: Patients will be treated as per department protocols and no additional intervention will be performed
Period: Overall Study
Arm/Group | All Participants
Started | 26
Completed | 26
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.58 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 26
Region of Enrollment [Number; unit: participants]
  Singapore | 26

OUTCOME MEASURES:

1. Primary Outcome: Degree of Disagreement, %
Description: Comparison of cardiac output monitoring capabilities of the NICOM Cheetah® versus the FloTrac®. Cardiac output defined as the amount of blood the heart pumps through the circulatory system in a minute. Bland-Altman analysis used to compare the level of disagreement between the 2 devices, %.
Time Frame: 10 hours of data collected for each participant
Measure: Number; unit: percentage of disagreement
Arm/Group | All Participants
Number analyzed (Participants) | 26
percentage of disagreement | 69.2

ADVERSE EVENTS:
Time Frame: 2 years
Description: All-Cause Mortality, Serious, or Other (non-serious) Adverse Events were monitored/assessed, but none observed.
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/26
Serious Adverse Events (participants affected / at risk) | 0/26
Other Adverse Events (participants affected / at risk) | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-24): https://cdn.clinicaltrials.gov/large-docs/68/NCT03394768/Prot_SAP_000.pdf